CLINICAL TRIAL: NCT00006427
Title: Management of Chronic Pain in Rehabilitation Project II Management of Chronic Pain in Persons With Amputation
Brief Title: Chronic Pain After Amputation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NICHD-0121; P01HD033988 (NIH)
Record Dates: First submitted 2000-11-01; First posted 2000-11-02 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2011-05

CONDITIONS: Amputation, Traumatic; Pain; Postoperative Pain
Keywords: Amputation; Chronic Pain; Amitriptyline
MeSH Terms: conditions — Amputation, Traumatic; Pain; Pain, Postoperative; Chronic Pain | interventions — Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline

SUMMARY:
This trial will test the effectiveness of amitriptyline in relieving chronic pain of adults that have had an amputation

DETAILED DESCRIPTION:
This double-masked placebo controlled trial will randomize patients (n=125) who are 6 months or more after amputation and have a 3 or more month history of pain to a daily dose of amitriptyline or a placebo for 6 weeks. Patients will receive a complete functional neurological examination by one of the study physicians or nurses masked to their treatment assignment. Study participants will also be interviewed by telephone to assess pain, pain interference with activities, physical and mental health, and number of health care visits for pain, at the beginning and end of the six-week trial and four months later.

ELIGIBILITY:
Inclusion Criteria:

* Amputation six months ago or longer
* Pain for 3 months or longer

Exclusion Criteria:

* History of cardiovascular disease, seizures, or glaucoma
* Currently taking antidepressant medications
* Currently hyperthyroid or taking thyroid medication
* Currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 1996-08; Primary Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Robinson, MD, Professor, Principal Investigator — University of Washington, Department of Rehabilitation
Locations (1):
- University of Washington, Department of Rehabilitation Medicine, Seattle, Washington, United States

REFERENCES:
- [Background] Davis RW. Successful treatment for phantom pain. Orthopedics. 1993 Jun;16(6):691-5. doi: 10.3928/0147-7447-19930601-10. PMID 8321759
- [Background] Onghena P, Van Houdenhove B. Antidepressant-induced analgesia in chronic non-malignant pain: a meta-analysis of 39 placebo-controlled studies. Pain. 1992 May;49(2):205-219. doi: 10.1016/0304-3959(92)90144-Z. PMID 1535121
- [Background] Philipp M, Fickinger M. Psychotropic drugs in the management of chronic pain syndromes. Pharmacopsychiatry. 1993 Nov;26(6):221-34. doi: 10.1055/s-2007-1014359. PMID 8127926
- See also: University of Washington, Department of Rehabilitation Medicine, Chronic Pain Study Website — http://depts.washington.edu/rehab/research/chronic.html
- See also: Click here for more information about the National Institute of Child Health and Human Development (NICHD). — http://www.nichd.nih.gov/